CLINICAL TRIAL: NCT02210715
Title: Randomized Study Comparing Switching to Raltegravir-based Antiretroviral Versus Maintaining Any Other Antiretroviral Therapy in HIV Monoinfected Patients Impact on Fatty Liver and Liver Fibrosis Assessed by Noninvasive Diagnostic Methods
Brief Title: Raltegravir-based Antiretroviral Versus Maintaining Any Other Antiretroviral Therapy in HIV Mono-infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Giada Sebastiani, Dr Giada Sebastiani MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: switchMerck
Record Dates: First submitted 2014-08-05; First posted 2014-08-07 (Estimated); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: HIV; Fatty Liver; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- switch to Isentress (Experimental): 28 subjects will be prescribed Raltegravir at the standard dose of 400 mg p.o. b.i.d. for 24 months.
  Interventions: Drug: Isentress.
- Continue usual antiretroviral therapy (Active Comparator): 28 subjects will continue with their normal cART treatment, as prescribed by their treating physician.
  Interventions: Other: Continue usual antiretroviral therapy

INTERVENTIONS:
Drug: Isentress. — 28 subjects will change from their normal cART treatment to Raltegravir, which will be given at the standard dose of 400 mg p.o. b.i.d. for 24 months.
  Other Names: Raltegravir
  Arms: switch to Isentress
Other: Continue usual antiretroviral therapy — 28 subjects will continue with their normal cART treatment, as prescribed by their treating physician.
  Arms: Continue usual antiretroviral therapy

SUMMARY:
People infected with HIV are living longer thanks to the use of antiretroviral therapy (cART). In aging HIV persons, other factors are associated with early death. One of the major factors is liver disease, which can be due to liver infections or reasons such as fatty liver. Fatty liver in the general population is a serious problem, affecting 30% of Canadian population. A specific type of fatty liver characterized by much inflammation, named nonalcoholic steatohepatitis (NASH) can lead to cirrhosis and death. Persons living with HIV can be at increased risk of NASH because of toxic effect of certain types of cART on the liver, obesity and other metabolic factors (for example diabetes). Some scientific data suggest that newer cART are associated with less fatty liver and liver damage. However, NASH has not been studied in detail in persons living with HIV. One reason for the lack of research is one of the only ways to detect liver disease is to undergo liver biopsy which can be painful and has complications. Recently, a new non-invasive technology (Fibroscan) has been developed which can tell doctors how much a liver is damaged and how much fat it contains without pain or complications. Moreover, a simple test measuring a specific protein in the blood, the cytokeratin 18 (CK-18), can help the diagnosis of NASH. We will study the effect of switching cART to newer types of HIV medication in patients with a non-invasive diagnosis of NASH done by Fibroscan and cytokeratin 18. We expect that switching older cART to less hepatotoxic drugs will lead to improvement of liver damage, fatty liver and NASH diagnosed by Fibroscan and cytokeratin 18. To evaluate this approach we plan to recruit 58 consenting HIV mono infected patients with non-invasive diagnosis of NASH and/or fatty liver with liver damage. Participants will undergo Fibroscan, a blood test for cytokeratin 18, a complete physical examination and laboratory tests every 3 months for 12 months, then at 18 and 24 months. The effect of the switching of HIV medications will be recorded. We anticipate that the current study will provide evidence for reduction of inflammation and liver damage with newer cART for treatment of HIV infection.

DETAILED DESCRIPTION:
Current Non-invasive tools for liver fibrosis and fatty liver/NASH, including Fibroscan/CAP and serum cytokeratin 18 (CK-18), are accurate and ideal for screening and monitoring. To date, there has been no study using these accurate non-invasive tools to prospectively evaluate the effect of switching cART to raltegravir in HIV mono-infected patients with suppressed HIV RNA who have evidence of fatty liver and/or significant liver fibrosis in order to determine whether such a strategy may slow fibrosis and steatosis progression rates.

Once a candidate for screening has been identified, study details will be carefully discussed with the subject. The subject will be asked to read and sign the approved informed consent form prior to any assessments being performed. Self-administered questionnaires will collect information on Alcohol use and Disorders Identification Test (audit C), drug use. chart review, (demographics, medication medical history).

Blood samples will be obtained for clinical laboratory evaluations (as per standard of care) at baseline, and all follow-up visits, plus serum CK-18 that will be obtained at all follow-up visits. Routine hematology and chemistry evaluations will include: complete blood count (CBC) with differential, CD4 and CD8 cell counts, viral load, C-reactive Protein, D-dimer, and measurements of hepatic, pancreatic and renal function, fasting insulin, creatine kinase, glucose and lipid profiles. Plasma HIV RNA levels will be measured with a lower limit of detection of 50 copies/mL. Clinical laboratory evaluations for hematology, biochemistry, CD4/CD8, viral load and serology will be performed at the chest institute as per local practices. Fibroscan will be performed on a fasting patient. The probe transducer will be placed on the skin, between the rib bones at the level of the right lobe of the liver. An experienced operator (> 500 examinations before the study), will perform the Fibroscan and the software will calculate the median . The standard M probe will be used in all patients. The XL probe will be used in obese patients (BMI>30 Kg/m2) or if the M probe fails to provide accurate results. CAP examination will be performed at the same time to diagnose fatty liver. A valid Fibroscan result will be defined by 10 validated measures and IQR < 30% of the median. The following cut-off values will be applied to diagnose fibrosis by Fibroscan: 1) 8 kilopascal (kPa) for significant liver fibrosis; 2) 13 kPa for cirrhosis. Fatty liver by CAP will be diagnosed with the following cut-off values: 1) 237.8 dB/m for mild steatosis; 2) 260 dB/m for moderate steatosis; 3) 292.3 dB/m for severe steatosis.

Subject Identification (ID) numbers will be assigned sequentially to each subject who is eligible to participate in the study. The Subject ID Number will consist of a three digit centre number and a three digit number according to chronological order of entry. If a patient discontinues from the study the Subject ID Number will not be reused. The Subject ID Numbers will be used for identification of subjects in the source documentation, and laboratory samples. This will ensure that subject data and laboratory samples leaving the study sites will be identified and tracked.

Randomization to study groups will be done using a computer-generated random allocation with stratification by gender. Summary statistics (mean, median, standard deviation, interquartile range) will be obtained for clinical and demographic data collected between baseline and study conclusion. The fatty liver and liver fibrosis scores by CAP and Fibroscan, respectively, at month 24 will be expressed as a function of exposure group, adjusting for baseline values of each outcome using an analysis of covariance (ANCOVA) model. The average difference in change of steatosis and fibrosis scores between the two groups and associated hypothesis tests will be obtained from the ANCOVA model. All analyses will be based on an intention-to-treat basis, that is, patients' data will be analyzed as randomized. To assess the sensitivity of inferences to missing data, we will generate plausible values for missing observations using multiple imputations (MI), which is a relatively objective methodology for handling missing data in longitudinal studies. In MI, multiple plausible values are generated for each missing item from the joint distribution of observed data using a Bayesian framework, and the results are pooled using established rules while simultaneously accounting for uncertainty in the imputation process. Multivariate logistic regression analysis will be used to explore factors associated with non-invasive diagnosis of fatty liver/NASH and significant liver fibrosis, including patient-related (age, gender, BMI), drug-induced (time on and type of cART), metabolic (diabetes, insulin resistance, lipid profile, hypertension), HIV-related (HIV viral load, CD4/CD8). Pearson correlation coefficient will be used to measure the association between CK-18 and Fibroscan/CAP values, BMI, transaminases. All hypotheses tests will be conducted at 5% level of significance (2-sided). Analyses will be performed using R program for Windows Release 2.13.1.

The trial will be monitored for safety and efficacy by a Data Safety Monitoring Board (DSMB) composed of clinicians, statisticians/methodologists and a lay member appointed by the McGill University Health center.

Adverse events (AEs) are defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the study medication/intervention. An AE can therefore be any unfavourable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug/intervention, whether or not it is related to the medication/intervention.

Stable chronic conditions which are present prior to clinical study entry and do not worsen are not considered adverse events and will be accounted for in the subject's medical history.

Subjects who have an adverse event should be followed and treated by the Investigator until the abnormal parameter or symptom has resolved or stabilized. It is up to the clinician to determine that the AE is either resolved or that is has reached a stable state, after which no further follow-up is necessary. There should also be source documentation to support this determination. At each contact with the subject, information regarding adverse events will be elicited by appropriate questioning and examinations, and will be recorded immediately on a source document (e.g., progress notes, laboratory reports, survey tools, and data collection tools). The start date, stop date, severity of each reportable event, and the PI's judgment of the AE's relationship to the study, medication/intervention will also be recorded.

Any AE that occurs between baseline and 30 days following Week 24 (or at the time of early discontinuation of the subject from the study for any reason) is to be recorded in the source documentation (patient will be called). Surveillance for AEs will end at 30 days following Week 24. If an serious adverse event (SAE) is ongoing at the time a subject discontinues/completes the trial the SAE will be followed until the Investigator agrees that the event is satisfactorily resolved or that no further follow-up is required.

Virologic failure must be considered for any patient with plasma HIV RNA ≥50 c/mL at any time following randomization. For the purposes of clinical management in this study, virologic failure is defined as: Two consecutive plasma HIV RNA ≥50 c/mL within four weeks of the initial suspected virologic failure. Cases of confirmed virologic failure will trigger genotypic virologic resistance testing, including integrase resistance testing, when plasma HIV RNA >400c/mL. The virologic failure definition is intended for guidance and Investigators should use their discretion as to the most appropriate clinical management of their patients. Due to the risk of developing integrase resistance in the setting of replicating HIV, change of antiretroviral therapy for subjects randomized to raltegravir is indicated for those with confirmed virologic failure. The choice of antiretroviral therapy will be left to the discretion of the treating physician.

The conduct of this study will conform to the International Conference for Harmonization and Good Clinical Practice (ICH-GCP) regulations and guidelines and the current revision of the Declaration of Helsinki A copy of the protocol (including protocol amendments), all versions of the informed consents, other information to be completed by subjects such as questionnaires, and any proposed advertising/ recruitment materials must be reviewed and approved by the research ethics board (REB) of each participating centre prior to implementation of the study. The investigator will be responsible for obtaining REB approval of the annual Continuing Review throughout the duration of the study. The investigator will notify the REB of violations from the protocol and SAEs.

All subjects will be given detailed oral and written information about the study. Consent forms describing in detail the study medications/intervention(s), study procedures, anticipated benefits and potential risks will be given to each participant and written documentation of informed consent is required prior to starting the study. Subjects must voluntarily sign and date an informed consent document that has been approved by the REB prior to any procedures being done specifically for the trial. Each subject should have sufficient opportunity to discuss the study and consider the information in the consent process prior to agreeing to participate. Subjects may withdraw consent at any time during the course of the trial. The informed consent will be signed and dated by the subject, the person who conducted the informed consent discussion and the investigator. The original signed informed consent form will be retained in the subject's study files and a copy will be provided to the subject.

All subject related information including the case report forms (CRFs), laboratory samples, evaluation forms, reports, etc. will be kept strictly confidential. All records will be kept in a secure, locked location and only research staff will have access to the records. Subjects will be identified only by means of a coded number specific to each subject, and a subject letter code. All computerized databases will identify subjects by numeric codes only, and will be password protected. Upon request, clinical information may be reviewed by or released to study monitors, auditors, Canadian Institutes of Health Research or regulatory agencies. The REB or other government organizations, as part of their duties to ensure that research subjects are protected may discontinue the study at any time. Regulatory authorities and the study Sponsor retain the authority to suspend additional enrollment for the entire study as applicable.

Data and study documents at all sites will be stored securely for 25 years, after which they will be destroyed in keeping with the privacy and confidentiality regulations and guidelines.

Appropriate medical and research records for this study and regulatory/ institutional requirements must be maintained for the protection of confidentiality of study subjects. The Principal Investigator is responsible for assuring that the data collected are complete, accurate, and recorded in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Confirmed positive serology for HIV mono-infection
3. Valid Fibroscan/CAP results
4. Able to provide informed consent (available in French or English)
5. Receiving any approved antiretroviral regimen that does not contain integrase-inhibitor
6. Evidence of fatty liver (CAP>237.8dB/m) AND/OR evidence of significant liver fibrosis (Fibroscan > 8KPa)
7. HIV viral suppression (<50 copies/mL) for at least 6 months
8. No prior evidence of resistance to raltegravir or co-administered nucleoside backbone

Exclusion Criteria:

1. Clinical evidence of decompensated liver disease at entry (e.g. ascites, bleeding esophageal varices, hepatic encephalopathy, or hepatoma/ hepatocellular carcinoma).
2. Co-infection with hepatitis C virus (HCV) or hepatitis C virus (HBV) (presence of serum HCV-Ab or HBsAg);
3. Alpha-fetoprotein (AFP) greater than or equal to 200 ng/mL at screening.
4. Known or suspected Wilson's disease, alpha-1-antitrypsin deficiency, celiac disease or other cause of chronic liver disease.
5. Chronic renal insufficiency (eGFR < 20 mL/min) at screening.
6. Pregnancy and planned pregnancy (not using adequate contraception).
7. Women who are breastfeeding.
8. Active opportunistic infection (except oral thrush) or neoplasm (except Kaposi's sarcoma, skin cancer, or cancer of the cervix or anus, unless known or suspected liver metastasis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-03; Primary Completion 2019-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
improvement of fatty liver or liver fibrosis | 24 months
  Difference in Fibroscan/CAP measurement from baseline to 24 months

SECONDARY OUTCOMES:
Difference in serum CK-18 levels | 24 months
  Difference in serum CK-18 levels as surrogate diagnostic marker of NASH from baseline to 24 months.
Difference in transaminases levels | 24 months
  Difference in transaminases levels (AST and/or ALT) from baseline to 24 months
Difference in metabolic markers | 24 months
  Difference in metabolic markers (HOMA; cholesterol or triglycerides levels; BMI) from baseline to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Giada Sebastiani, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada